CLINICAL TRIAL: NCT06172959
Title: The Short-term Impact of Vocal Intonation Therapy (VIT) and Therapeutic Singing (TS) on Respiratory Function in Patients With Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Teresa Lesiuk, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20230944
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vocal Therapy Group (Experimental): Participants in this group will receive Vocal Intonation Therapy (VIT) and Therapeutic Singing (TS) for up to three weeks
  Interventions: Behavioral: Vocal Intonation Therapy (VIT); Behavioral: Therapeutic Singing (TS)

INTERVENTIONS:
Behavioral: Vocal Intonation Therapy (VIT) — Participants will receive 12 individual sessions, four times a week (i.e., any four days of seven days) over three weeks. Each session will be held virtually for 30-minutes. Vocal Intonation Therapy is a music therapy technique consisting of breathing and vocal exercises to target respiratory function and vocal quality.
Behavioral: Therapeutic Singing (TS) — Participants will receive 12 individual sessions, four times a week (i.e., any four days of seven days) over three weeks. Each session will be held virtually for 30-minutes. Therapeutic Singing is a music therapy technique used to work on the rehabilitation of vocal and respiratory function.

SUMMARY:
The purpose of this study is to examine the short-term impact of Vocal Intonation Therapy (VIT) and Therapeutic Singing (TS) on respiratory function in patients with lung cancer. As a secondary outcome, this research will evaluate the effect of the music intervention on respiratory quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Participants will include three patients diagnosed with lung cancer, stages I-III, who have undergone a thoracentesis or thoracotomy in the last 12 months. Thoracic surgical procedures include pulmonary lobectomy or cancer-related surgical procedure (e.g., pneumonectomy). This diagnosis must be made by the patient's oncologist and medical team.
* The age range will be 40 to 80 years old. Both female and male participants from any race and ethnicity will be included in the study.
* The study will include English and Spanish speakers only.
* Patients must have less than five years of voice training experience (e.g., choir, private voice lessons).

Exclusion Criteria:

* Patients in respiratory failure
* Individuals with severe neurological and hearing impairments.
* Patients with diagnosed dysphonia and individuals who have undergone a laryngectomy
* Participants that do not have access to an electronic device, either an iPad, tablet, or laptop, as well as reliable internet access. They will also need to have adequate knowledge of technology or participate with a caregiver who knows how to navigate Zoom.
* Participants who do not have access to a quiet space. Headphones are optional for this study.
* Prisoners
* Persons under the age of 40 or over the age of 80.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Maximum Phonation Time (MPT) in seconds | Baseline, up to 30-minutes (Post-Intervention)
  Maximum Phonation Time (MPT) measures the number of seconds a participant can sustain a phonated sound.
Respiratory Rate | Up to 30-minutes
  Measured by the number of breaths per minute
Change in Dyspnea measured by Dyspnea-12 Questionnaire | Baseline, up to 1 month
  Scores range from 0 to 3. Higher scores suggest more severity in shortness of breath
Change in Dyspnea measured by Modified Borg Scale | Baseline, up to 30-minutes (Post-Intervention)
  Scores change from 0 to 10. Higher scores suggest more severity in shortness of breath
Change in Respiratory Quality of Life measured by St.Georges Respiratory Questionnaire | Baseline, up to 1 month
  A composite score will be obtained, ranging from 0 to 100. Higher scores indicate worst respiratory quality of life
Change in Dyspnea measured by Cancer Dyspnea Scale | Baseline, up to 1 month
  Scores range from 1 (Not at all) to 5 (Very much). Higher scores suggest more severity of dyspnea

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Lesiuk, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No